CLINICAL TRIAL: NCT06915558
Title: Modulation of the Inflammatory Response to Surgical Trauma: Comparison of Three Anesthetic Techniques in Bariatric Surgery Patients
Brief Title: Modulation of the Inflammatory Response in Bariatric Surgery
Acronym: MRICBx3
Status: Recruiting | Type: Observational
Sponsor: Hospital HM Nou Delfos (Other)
Responsible Party: Principal Investigator, HIPÓLITO LABANDEYRA GONZALEZ, Anesthesiologist, Hospital HM Nou Delfos
Other Study IDs: 25.02.2467-GHM
Record Dates: First submitted 2025-03-24; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Obesity; Bariatric Surgery Candidate; Inflammation; Postoperative Pain; Opioid-Free Anesthesia; Heart Rate Variability
Keywords: Opioid-Free Anesthesia; Opioid-Based Anesthesia; Inflammatory Markers; Surgical Stress Response; heart rate variability
MeSH Terms: conditions — Obesity; Inflammation; Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Opioid-Free Anesthesia (OFA): Patients in this group will receive opioid-free anesthesia (OFA) using a multimodal analgesic approach, including dexmedetomidine, lidocaine, ketamine, and magnesium sulfate. No intraoperative opioids will be administered. Inflammatory biomarkers (IL-6, PCR, cortisol, WBC, VSG) and heart rate variability (HRV) will be measured to assess the inflammatory response.
  Interventions: Procedure: Opioid-Free Anesthesia (OFA)
- Opioid-Based Anesthesia - Intravenous (OBA-IV): Patients in this group will receive opioid-based intravenous anesthesia (OBA-IV) with propofol, remifentanil, and neuromuscular blockade. Standard opioid-based analgesia will be administered intraoperatively. Inflammatory biomarkers (IL-6, PCR, cortisol, WBC, VSG) and HRV will be assessed to compare inflammatory responses between opioid-based and opioid-free techniques.
  Interventions: Procedure: Opioid-Based Intravenous Anesthesia (OBA-IV)
- Opioid-Based Anesthesia - Inhalational (OBA-Inh): Patients in this group will receive opioid-based inhalational anesthesia (OBA-Inh) using sevoflurane, remifentanil, and neuromuscular blockade. Standard opioid-based analgesia will be used intraoperatively. Inflammatory biomarkers (IL-6, PCR, cortisol, WBC, VSG) and HRV will be analyzed to evaluate differences in the inflammatory response among the three anesthetic techniques.
  Interventions: Procedure: Opioid-Based Inhalational Anesthesia (OBA-Inh)

INTERVENTIONS:
Procedure: Opioid-Free Anesthesia (OFA) — Opioid-free anesthesia using a multimodal approach, including dexmedetomidine, lidocaine, ketamine, and magnesium sulfate. No intraoperative opioids are administered.
  Other Names: Multimodal Opioid-Free Anesthesia
  Groups: Opioid-Free Anesthesia (OFA)
Procedure: Opioid-Based Intravenous Anesthesia (OBA-IV) — Standard opioid-based intravenous anesthesia using propofol, remifentanil, and neuromuscular blockade.
  Other Names: IV Opioid-Based Anesthesia
  Groups: Opioid-Based Anesthesia - Intravenous (OBA-IV)
Procedure: Opioid-Based Inhalational Anesthesia (OBA-Inh) — Standard opioid-based inhalational anesthesia using sevoflurane, remifentanil, and neuromuscular blockade.
  Other Names: Inhalational Opioid-Based Anesthesia
  Groups: Opioid-Based Anesthesia - Inhalational (OBA-Inh)

SUMMARY:
This study will evaluate how different anesthesia techniques affect inflammation after bariatric surgery. Patients will be randomly assigned to receive one of three approaches: opioid-free anesthesia, intravenous anesthesia with opioids, or inhalational anesthesia with opioids.

The study will measure blood levels of inflammation-related substances (such as IL-6, CRP, cortisol, ESR , WBC and lactate) at several time points before and after surgery. Heart rate variability will also be monitored as an indicator of the body's stress response.

The results may help identify anesthesia strategies that reduce inflammation and improve recovery in patients undergoing bariatric surgery.

DETAILED DESCRIPTION:
This is a prospective, randomized, double-blind, comparative observational study designed to assess the perioperative inflammatory response in patients undergoing bariatric surgery under three anesthetic techniques: opioid-free anesthesia (OFA), opioid-based intravenous anesthesia (OBA-IV), and opioid-based inhalational anesthesia (OBA-Inh).

A total of 90 patients scheduled for elective laparoscopic bariatric surgery will be enrolled and randomized using computer-generated allocation into three equal groups (n=30 each). Allocation concealment will be maintained using sealed opaque envelopes. Blinding will involve both the patients and outcome assessors; anesthesiologists administering the interventions will not be blinded due to the nature of the techniques.

The study's primary focus is to evaluate the perioperative modulation of inflammation through quantification of biomarkers including interleukin-6 (IL-6), C-reactive protein (CRP), serum cortisol, leukocyte count (WBC), erythrocyte sedimentation rate (ESR) and lactate. Heart rate variability (HRV) will be continuously monitored as a surrogate marker for autonomic modulation of the inflammatory response.

Biomarkers will be sampled at three time points: preoperative baseline (T0), at the end of surgery (T1), and 24 hours postoperatively (T2). HRV data will be collected from induction to the end of surgical intervention using a non invasive monitoring system with time- and frequency-domain analysis.

Secondary outcomes include intraoperative and postoperative analgesic consumption, pain intensity assessed by visual analog scale (VAS), sedation scores using the Ramsay Agitation-Sedation Scale (RASS), incidence of opioid-related side effects (nausea, vomiting, respiratory depression), patient satisfaction (via validated questionnaire), and length of hospital stay.

Sample size was calculated based on preliminary data detecting a clinically significant difference in IL-6 levels, assuming an alpha of 0.05 and power of 0.8. Data will be analyzed using ANOVA or Kruskal-Wallis test for continuous variables, chi-square for categorical variables, and multivariate regression models to adjust for potential confounders.

This study aims to identify anesthetic strategies that minimize systemic inflammation and autonomic dysregulation in the bariatric surgical population, with potential applications in broader surgical settings.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for bariatric surgery.
* Age 18-65 years.
* BMI ≥ 30 kg/m².
* ASA physical status II-III.

Exclusion Criteria:

* Pregnancy or breastfeeding.
* Chronic opioid use before surgery.
* Severe renal or hepatic failure.
* Uncontrolled psychiatric disorders.
* Significant intraoperative complications requiring protocol deviation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients undergoing elective bariatric surgery at HM Nou Delfos Hospital. Patients will be selected according to specific inclusion and exclusion criteria to ensure homogeneous groups for the comparison of inflammatory response to different anesthetic techniques. All participants will undergo preoperative screening, intraoperative monitoring, and postoperative follow-up to evaluate primary and secondary outcomes.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2025-12-02 (Estimated); Study Completion 2025-12-02 (Estimated)

PRIMARY OUTCOMES:
Serum IL-6 Level | Preoperative (baseline), immediately after surgery, and 24 hours post-surgery.
  Measurement of interleukin-6 (IL-6) concentration in pg/mL to evaluate inflammatory response.
C-reactive Protein (CRP) Level | Preoperative (baseline), immediately after surgery, and 24 hours post-surgery.
  Measurement in mg/L to assess systemic inflammation.
Serum Cortisol Level | Preoperative (baseline), immediately after surgery, and 24 hours post-surgery.
  Measurement in μg/dL.
Heart Rate Variability (HRV) as an Inflammatory Marker | Collected continuosly from the induction of the anesthesia until the end of surgery
  Heart Rate Variability (HRV) as an Inflammatory Marker and its correlation with blood levels of inflammatory markers Heart Rate Variability (HRV) as an Indicator of Inflammatory Response
Serum Lactate Level | Preoperative (baseline), immediately after surgery, and 24 hours post-surgery.
  Measurement in mmol/L as a marker of metabolic response.
Erythrocyte Sedimentation Rate (ESR) | Preoperative (baseline), immediately after surgery, and 24 hours post-surgery.
  Measurement of ESR in mm/h to assess systemic inflammation.
Differential White blood Cell count (WBC). | Preoperative (baseline), immediately after surgery, and 24 hours post-surgery.
  Measurement of total white blood cell count in peripheral blood, expressed in thousands of cells per microliter (10³/μL). Assessment of the percentage distribution of white blood cell subtypes, including neutrophils, lymphocytes, monocytes, eosinophils, and basophils, expressed as a percentage of total leukocytes.

SECONDARY OUTCOMES:
Postoperative Pain Evaluation Using Visual Analog Scale (VAS) | hourly during the first 4 hours post surgery in the recovery area, and at 12 and 24 hours in the hospitalization ward
  Assessment of pain intensity using the Visual Analog Scale (VAS), a 10 cm scale ranging from 0 (no pain) to 10 (worst imaginable pain). Higher scores indicate greater pain intensity.
Postoperative Sedation Level Using Ramsay Sedation Scale | immediately after surgery, and hourly during the first 4 hours in the recovery area, and at 12 and 24 hours in the hospitalization ward
  Evaluation of sedation using the Ramsay Sedation Scale, which ranges from 1 (anxious and agitated) to 6 (no response to stimulus). Higher scores indicate deeper levels of sedation.
Incidence of Postoperative Complications | 24 hours post-surgery.
  Measurement of total hospital stay (in days) after surgery.
Patient Satisfaction with Anesthetic Technique | 24 hours post-surgery.
  Evaluation of patient satisfaction using a standardized 5-point Likert scale questionnaire (1 = very dissatisfied; 5 = very satisfied) regarding anesthesia and overall recovery experience.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Contreras-Pérez, Anesthesiologist, Principal Investigator — Hospital HM Nou Delfos
Locations (1):
- Hospital HM Nou Delfos, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to privacy regulations and ethical considerations. Data will only be accessible to the research team and authorized personnel as per institutional and regulatory guidelines.

REFERENCES:
- [Background] Heil LBB, Silva PL, Pelosi P, Rocco PRM. Immunomodulatory effects of anesthetics in obese patients. World J Crit Care Med. 2017 Aug 4;6(3):140-152. doi: 10.5492/wjccm.v6.i3.140. eCollection 2017 Aug 4. PMID 28828299
- [Background] Alsumali A, Eguale T, Bairdain S, Samnaliev M. Cost-Effectiveness Analysis of Bariatric Surgery for Morbid Obesity. Obes Surg. 2018 Aug;28(8):2203-2214. doi: 10.1007/s11695-017-3100-0. PMID 29335933
- [Background] Lin YT, Wu HT, Tsao J, Yien HW, Hseu SS. Time-varying spectral analysis revealing differential effects of sevoflurane anaesthesia: non-rhythmic-to-rhythmic ratio. Acta Anaesthesiol Scand. 2014 Feb;58(2):157-67. doi: 10.1111/aas.12251. PMID 24410106
- [Background] Bonhomme V, Uutela K, Hans G, Maquoi I, Born JD, Brichant JF, Lamy M, Hans P. Comparison of the surgical Pleth Index with haemodynamic variables to assess nociception-anti-nociception balance during general anaesthesia. Br J Anaesth. 2011 Jan;106(1):101-11. doi: 10.1093/bja/aeq291. Epub 2010 Nov 4. PMID 21051493
- [Background] Wennervirta J, Hynynen M, Koivusalo AM, Uutela K, Huiku M, Vakkuri A. Surgical stress index as a measure of nociception/antinociception balance during general anesthesia. Acta Anaesthesiol Scand. 2008 Sep;52(8):1038-45. doi: 10.1111/j.1399-6576.2008.01687.x. PMID 18840101
- [Background] Lisowska B, Jakubiak J, Siewruk K, Sady M, Kosson D. Which idea is better with regard to immune response? Opioid anesthesia or opioid free anesthesia. J Inflamm Res. 2020 Nov 5;13:859-869. doi: 10.2147/JIR.S275986. eCollection 2020. PMID 33177861
- [Background] Campos-Perez W, Ramirez-Plascencia L, Perez-Robles M, Rivera-Valdes JJ, Sanchez-Munoz P, Perez-Vargas L, Gonzalez-Landeros D, Cuevas JHM, Martinez-Lopez E. A comparison of opioid-containing anesthesia versus opioid-free anesthesia using the Cortinez-Sepulveda model on differential cytokine responses in obese patients undergoing gastric bypass surgery: a randomized controlled trial. BMC Anesthesiol. 2022 Sep 16;22(1):294. doi: 10.1186/s12871-022-01838-8. PMID 36114460
- [Background] Ahmed SA, Abdelghany MS, Afandy ME. The effect of opioid-free anesthesia on the post-operative opioid consumption in laparoscopic bariatric surgeries: A randomized controlled double-blind study. J Opioid Manag. 2022 Jan-Feb;18(1):47-56. doi: 10.5055/jom.2022.0694. PMID 35238013
- [Background] Schneemilch CE, Ittenson A, Ansorge S, Hachenberg T, Bank U. Effect of 2 anesthetic techniques on the postoperative proinflammatory and anti-inflammatory cytokine response and cellular immune function to minor surgery. J Clin Anesth. 2005 Nov;17(7):517-27. doi: 10.1016/j.jclinane.2004.12.017. PMID 16297751
- [Background] Lin E, Calvano SE, Lowry SF. Inflammatory cytokines and cell response in surgery. Surgery. 2000 Feb;127(2):117-26. doi: 10.1067/msy.2000.101584. PMID 10686974
- [Background] Schumann R. Anaesthesia for bariatric surgery. Best Pract Res Clin Anaesthesiol. 2011 Mar;25(1):83-93. doi: 10.1016/j.bpa.2010.12.006. PMID 21516916
- [Background] Ellulu MS, Patimah I, Khaza'ai H, Rahmat A, Abed Y. Obesity and inflammation: the linking mechanism and the complications. Arch Med Sci. 2017 Jun;13(4):851-863. doi: 10.5114/aoms.2016.58928. Epub 2016 Mar 31. PMID 28721154
- [Background] Gregor MF, Hotamisligil GS. Inflammatory mechanisms in obesity. Annu Rev Immunol. 2011;29:415-45. doi: 10.1146/annurev-immunol-031210-101322. PMID 21219177